CLINICAL TRIAL: NCT05669950
Title: A Multi-site, Open-label, Sequential-group, Multiple-dose Trial to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamic Effects of Lu AG13909 in Participants With Congenital Adrenal Hyperplasia
Brief Title: A Trial of Lu AG13909 in Participants With Congenital Adrenal Hyperplasia
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 19873A
Record Dates: First submitted 2022-12-20; First posted 2023-01-03 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Congenital Adrenal Hyperplasia
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lu AG13909 (Experimental): Participants in Part A will receive multiple intravenous (IV) doses of Lu AG13909 per a prespecified dosing schedule. After data from Part A has shown that a pharmacologically relevant dose level is safe and tolerable, participants in Part B will then receive multiple IV doses of Lu AG13909 per a prespecified dosing schedule. After data from Part B has shown that a pharmacologically relevant dose level is safe and tolerable, participants in Part C will then receive multiple IV doses of Lu AG13909 per a prespecified dosing schedule. Participants from Part C may be eligible to continue in the optional Treatment Extension.
  Interventions: Drug: Lu AG13909

INTERVENTIONS:
Drug: Lu AG13909 — Solution for infusion

SUMMARY:
This trial will evaluate the effects of different doses of Lu AG13909 in adult participants with congenital adrenal hyperplasia, also called CAH. CAH is a rare genetic disorder that affects a person's ability to produce certain hormones. The main goals of this trial are to learn about the safety and tolerability of Lu AG13909, how Lu AG13909 behaves in the body, and how the body responds to Lu AG13909.

ELIGIBILITY:
Inclusion Criteria:

Parts A and B:

* Confirmed diagnosis of 21-hydroxylase deficiency CAH (based on a pathogenic CYP21A2 variant and/or elevated 17-OHP).
* Morning (pre-glucocorticoid [GC] replacement dose) blood concentrations of 17-OHP >4-times upper limit of normal (ULN).
* Body mass index (BMI) ≥18.5 kilograms (kg)/square meter (m^2) (minimum 50 kg) and ≤40 kg/m^2.
* Stable GC replacement therapy for ≥1 month prior to the Screening Visit.
* For the salt-wasting form of CAH, the participant must have been on a stable dose of mineralocorticoid replacement for ≥3 months prior to the Screening Visit.
* Apart from CAH, the participant is generally healthy in the opinion of the investigator and based on medical history, physical examination, vital signs, ECGs, and the results of the safety laboratory tests.

Part C:

* Confirmed diagnosis of 21-hydroxylase deficiency CAH (based on a pathogenic CYP21A2 variant and/or elevated 17-OHP).
* For Cohort C1 only: Morning (pre-GC replacement dose) blood concentrations of androgens (A4) > ULN for age and sex.
* For Cohort C2 only: Morning (pre-GC replacement dose) blood concentrations of androgens (A4) ≤ ULN for age and sex and the participant is treated with high doses of GC.
* Stable GC replacement therapy for ≥1 month prior to the Screening Visit.
* For the salt-wasting form of CAH, the participant must have been on a stable dose of mineralocorticoid replacement for ≥1 month prior to the Screening Visit.

Exclusion Criteria:

* The participant is pregnant or breastfeeding.
* The participant has a clinically significant abnormal laboratory value, electrocardiogram (ECG) parameter, or vital signs value, or other safety findings at the Screening Visit that indicate a potential risk for the participant if enrolled, in the opinion of the investigator.
* The participant has a history of known hypersensitivity or intolerance to Lu AG13909 or its excipients.

Part C Only:

* The participant has received at least one dose of Lu AG13909 in Part A or Part B.

Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-12-19 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Parts A and B: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) | Up to Day 161
Parts A and B: Number of Participants With Anti-Drug Antibodies (ADAs) | Day 1 up to Day 161
Parts A and B: Cmax: Maximum Observed Serum Concentration of Lu AG13909 | 0 (predose) up to 24 hours postdose on Day 1 to Day 161
Parts A and B: Tmax: Nominal Time Corresponding to the Occurrence of Cmax | 0 (predose) up to 24 hours postdose on Day 1 to Day 161
Parts A and B: Ctrough: Minimum Observed Serum Concentration of Lu AG13909 | 0 (predose) up to 24 hours postdose on Day 1 to Day 161
Parts A and B: t½: Apparent Elimination Half-life of Lu AG13909 | 0 (predose) up to 24 hours postdose on Day 1 to Day 161
Parts A and B: AUC0-infinity: Area under the plasma concentration curve of x from zero to infinity of Lu AG13909 | 0 (predose) up to 24 hours postdose on Day 1 to Day 161
Parts A and B: CL: Apparent Total Serum Clearance of Lu AG13909 | 0 (predose) up to 24 hours postdose on Day 1 to Day 161
Parts A and B: Vz: Volume of Distribution During the Terminal Elimination Phase After IV Administration of Lu AG13909 | 0 (predose) up to 24 hours postdose on Day 1 to Day 161
Parts A and B: Change From Baseline After Each Dose of Lu AG13909 in Blood Concentrations of 17-hydroxyprogesterone (17-OHP) and Androstenedione (A4) | Baseline up to Day 85
Parts A and B: AUC0-tau: Area under the curve over a dosing interval | 0 (predose) up to 24 hours postdose on Day 1 to Day 161
Part C: Morning Concentration of A4 in Blood <Upper Limit of Normal (ULN) | Day 169

SECONDARY OUTCOMES:
Part C: Lu AG13909 Serum Concentrations Following Multiple IV Doses | Baseline up to Day 352
Part C: Change From Baseline of Lu AG13909 in Blood Concentrations of 17-OHP and A4 | Baseline up to Day 169
Part C: Number of Participants With TEAEs | Baseline up to Day 352
Part C: Number of Participants With ADAs | Baseline up to Day 352

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — HQ_Medinfo@Lundbeck.com
Locations (8):
- Rigshospitalet, Copenhagen, Denmark
- GH Pitié-Salpêtrière, Paris, France
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg
  - Karolinska University Hospital, Stockholm
- United Kingdom (4):
  - NIHR/Wellcome Trust Clinical Research Facility, Birmingham
  - Cambridge Clinical Research Centre, Cambridge
  - NIHR Clinical Research Facility, London
  - University College London Hospital - NIHR, London